CLINICAL TRIAL: NCT00409084
Title: Beta Blockers Versus Variceal Band Ligation and Beta Blockers for Primary Prophylaxis of Variceal Bleeding
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Arun J. Sanyal, MD, Virginia Commonwealth University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM10546
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Esophageal Varices
Keywords: varices; band ligation; portal hypertension; primary prophylaxis; cirrhosis; beta blockers
MeSH Terms: conditions — Esophageal and Gastric Varices; Varicose Veins; Hypertension, Portal; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): endoscopic variceal band ligation
  Interventions: Procedure: endoscopic variceal band ligation
- 2 (Active Comparator): subjects will receive nadolol (beta blocker) at 20mg/day with dose titration
  Interventions: Procedure: endoscopic variceal band ligation

INTERVENTIONS:
Procedure: endoscopic variceal band ligation — endoscopic variceal band ligation

SUMMARY:
Patients with scarring of the liver (cirrhosis) and portal hypertension (elevated blood pressure in the liver vasculature) can develop esophageal varices (dilated veins). These have an increased risk of bleeding each year. Current recommendations are to prevent bleeding of medium or large varices (when there is no history of bleeding) by starting a blood pressure lowering agent known as a non-selective beta-blocker. Alternatively, rubber bands can be placed on medium to large varices to prevent bleeding (endoscopic variceal band ligation). Using both therapies at the same time has not been studied. In this study, we hope to determine if the use of combination therapy with endoscopic variceal band ligation and beta blockers is more effective than using beta blockers alone to prevent the first bleeding episode from the varices (dilated veins). The efficacy, ability to tolerate, and cost-effectiveness of these two treatment strategies will be compared.

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis
* medium to large varices

Exclusion Criteria:

* contraindications to beta blockers
* refusal to give consent
* prior history of variceal hemorrhage
* creatinine > 1.5 mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
first variceal bleed | 2 years

SECONDARY OUTCOMES:
survival | 2 years
liver function | 1 year
encephalopathy | 1 year
quality of life | 1 year
frequency of other complications of cirrhosis | 2 years
cost utility | 1 year
patient preference | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, M.D., Principal Investigator — Division of Gastroenterology, Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States